CLINICAL TRIAL: NCT02497430
Title: A Multi-Site Clinical Evaluation of the ARIES Group B Streptococcus (GBS) Assay With Vaginal-Rectal Swab Specimens From Antepartum Pregnant Women
Brief Title: Clinical Evaluation of the ARIES Group B Streptococcus (GBS) Assay
Status: Completed | Type: Observational
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-GBS-01-CS-001
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy; GBS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vaginal-rectal swab
Oversight: Data Monitoring Committee: No

SUMMARY:
The ARIES GBS Assay is a real-time PCR based qualitative test designed to detect Group B Streptococcus (GBS) nucleic acid from Lim Broth enriched vaginal-rectal specimen swabs obtained from pregnant women between 35 - 37 weeks gestation.

DETAILED DESCRIPTION:
The ARIES GBS Assay is a real-time polymerase chain reaction (PCR) based qualitative in vitro diagnostic test designed to detect Group B Streptococcus (GBS) nucleic acid from Lim Broth enriched vaginal-rectal specimen swabs obtained from pregnant women.

The objective of this study is to establish the diagnostic accuracy of ARIES GBS Assay through a multi-site, method comparison on prospectively collected, left-over enriched Lim broth specimens.

Diagnostic accuracy will be expressed in terms of clinical sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

1. An exemption from the requirement for Informed Consent has been granted by the site IRB to include the left-over patient specimens in the study.
2. Demographic information, including age, geographic location, and number of gestation weeks, is included with the specimen.
3. The specimen is from a female patient who is at 35 - 37 weeks gestation.
4. The specimen was collected in unexpired liquid Transport Media (e.g., Liquid Stuart or Liquid Amies).
5. Enrichment in Lim broth was grown for ≥18 hrs to ≤24 hrs.
6. The specimen is received in good condition (no leakage or drying of the specimen) and was accepted for testing by the site in accordance with established laboratory procedures.
7. The volume of the patient specimen after enrichment is sufficient (≥ 1.75mL) for completion of the study.

Exclusion Criteria:

1. The specimen was collected at a site which is not covered under the study IRB.
2. The specimen is from a patient for whom demographic data - age, geographic location and/or gestation weeks cannot be obtained.
3. The specimen was not properly collected, identified, transported, processed or stored according to the instructions provided by the Sponsor.
4. The specimen was enriched in Lim broth for <18 hrs or >24 hrs.
5. A swab specimen that cannot be placed in Lim broth within 4 days of collection.
6. Inconclusive latex agglutination results - weak agglutination, agglutination that occurs in more than one latex reagent or the results are otherwise considered inconclusive based on established laboratory procedures or the instructions included with the latex agglutination test kit.
7. Any specimen that was not tested per the complete testing algorithm provided by the Sponsor.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All comers
Sampling Method: Probability Sample
Enrollment: 918 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy expressed in terms of clinical sensitivity and clinical specificity | Within the first year of sample collection

SECONDARY OUTCOMES:
Comparison of clinical performance per clinical site and per age group | Within the first year of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Dunn, Study Director — Luminex Corporation
Locations (5):
- United States (5):
  - Sacred Heart Health System, Pensacola, Florida
  - Detroit Medical Center University Laboratories, Detroit, Michigan
  - TriCore Reference Laboratories, Albuquerque, New Mexico
  - Geisinger Medical Laboratories, Danville, Pennsylvania
  - Baylor Scott & White, Temple, Texas